CLINICAL TRIAL: NCT06375694
Title: Oral Probiotic Effect on Dietary Nitrate to Plasma Nitrite Production
Brief Title: Probiotic Effect on Dietary Nitrate to Plasma Nitrite Production ( OPEDNPN )
Acronym: OPEDNPN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University (Other)
Collaborators: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB00025485
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Hypertension; Cardiovascular Diseases; Diabetes
Keywords: Nitric Oxide; Nitrate; Microbiome
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into two groups with one group receiving the oral probiotic and the other receiving the placebo. Each group will take their intervention 2X a day for 7 days.
Who Masked: Participant
Masking Description: Participants will not know which group they are in. The lozenges will be distributed in unmarked bottles
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Active Comparator): Participants will take the commercially available oral probiotic (Herbiotics Oral + Ent Probiotic) twice a day for 7 days as instructed by the manufacturer. This entails one lozenge twice a day taken by mouth and slowly chewed or allowed to melt in the mouth.
  Interventions: Dietary Supplement: Herbiotics Oral + Ent Probiotic
- Placebo (Placebo Comparator): Participants will take the commercially available Honest Placebo Pills by Zeebo twice a day for 7 days. This entails one tablet twice a day taken by mouth and slowly chewed or allowed to melt in the mouth.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Herbiotics Oral + Ent Probiotic — Chewable Tablets containing Lactobacillus species.
  Arms: Probiotic
Dietary Supplement: Placebo — Honest Placebo Pills by Zeebo
  Arms: Placebo

SUMMARY:
Nitric Oxide (NO) is an important molecule that is produced naturally in the body and that helps maintain healthy blood flow. Low availability of NO contributes to many diseases while administration of NO is therapeutic.

In addition to being made naturally in the body, NO can be obtained through the diet via the Nitrate-Nitrite-NO cycle. Nitrate, which is abundant in green leafy vegetables and beetroot juice, is partially converted to nitrite by oral bacteria. The nitrate and nitrite are taken up into the blood and nitrite is converted into NO. Remaining nitrate in the blood is taken back up into the mouth by salivary glands and the cycle continues. Emerging studies suggest that the Nitrate-Nitrite-NO cycle may contribute to cardiovascular health. In addition, there have been many studies where dietary nitrate is given to increase NO and treat various conditions.

The current study rests on the premise that the quality of the oral microbiome plays a major role in the Nitrate-Nitrite-NO cycle and hence cardiovascular health and the efficacy of dietary nitrate interventions. Investigators have begun to identify oral bacterial species that are effective nitrite producers as well as though that are nitrite depleters (those that interfere with nitrite production from nitrate).

In laboratory experiments, certain bacterial species have been shown to block nitrate to nitrite conversion by other oral bacteria. These nitrite depleting species are found in a commercially available oral probiotic designed to improve oral health. The purpose of this study is to examine if use of the probiotic negatively affects the Nitrate-Nitrite-NO cycle. Nitrate to Nitrite conversion will be assessed by measuring plasma levels of nitrite before and after consumption of nitrate-rich beetroot juice. Dietary nitrate to plasma nitrite conversion will assessed at baseline and after one week of consumption of the probiotic or a placebo (follow-up). The primary hypothesis of this study is that participants that consume the probiotic will have lower nitrate to nitrite conversion at follow-up compared to baseline and that there will be no significant change in nitrate to nitrite conversion between baseline and follow-up for participants who consume the placebo.

While this study does not aim to treat any specific disease, it is intended to elucidate a basic physiological function that may be relevant to cardiovascular health and certain NO-based therapeutics.

DETAILED DESCRIPTION:
Background

Nitric oxide (NO) plays critical roles in a myriad of cellular and molecular mechanisms regulating physiology and function of various organs and systems.1,2 Low NO bioavailability contributes to pathology in multiple diseases including hemolytic anemias,3 malaria,4,5 transfusion of older stored blood,6,7 chronic heart failure,8 atherosclerosis,9 and diabetes.10 Recent reports suggest that the oral microbiome is linked with regulating NO homeostasis through the action of certain bacteria that have an ability to reduce nitrate to nitrite.11-15 Nitrite is then further reduced to NO through a variety of mechanisms in different tissues.16,17 Plasma nitrate is taken up back into the oral cavity by salivary glands so that the nitrate-nitrite-NO cycle provides sustained increases in NO bioavailability. Many clinical studies have used dietary nitrate as a source of NO through nitrite conversion.18-24 However, there is substantial variability in the clinical outcomes due to dietary nitrate intake and this is reflected in variability in the amount of nitrate converted to plasma nitrite.13,24-29 30. The variability and hence a large overall limitation in efficacy of dietary nitrate based treatments has been attributed to the capacity of the oral microbiome to reduce nitrate to nitrite.24-27 Preliminary work has begun to identify bacterial strains that are efficient nitrate to nitrite converters as well as those that actually inhibit nitrate to nitrite conversion.31,32 The efficiency of the nitrate-nitrite-NO cycle and the role of oral bacteria may contribute to normal health.11 Thus, understanding the variability in nitrate to nitrite conversion and aspects of the oral microbiome could lead to improvements in normal cardiovascular health. In addition, in order to maximize benefits from dietary nitrate interventions, we need to understand factors of the oral microbiome that affect nitrate to nitrite conversion. The investigators have recently discovered that several species of Lactobacillus produce a metabolite that blunts nitrate to nitrite conversion by other oral bacteria in vitro. Several of these Lactobacillus species are the main component of a commercially available oral probiotic, https://www.amazon.com/Dental-Probiotics-Breath-Gingivitis-Throat/dp/B096SZSFFS

Purpose

The purpose of this study is to determine if Lactobacillus will blunt dietary nitrate to plasma nitrite conversion.

The investigators hypothesize that the presence of oral Lactobacillus will blunt the conversion of dietary nitrate to plasma nitrite and will test this by comparing the conversion before and after use of this probiotic.

The main hypothesis rests on the auxiliary hypothesis that use of the oral probiotic will results in increased abundance of Lactobacillus in the oral cavity and will test this through genomic sequencing.

Methods OPEDNPN All eligible volunteers will be consented after learning about the study and agreeing to participate. Volunteers will be randomly assigned to one of two groups: (1) Probiotic and (2) Placebo. A total of 20 volunteers (10 per group) will participate in the study. The only difference for participants for each group will be whether they receive the placebo or probiotic.

All volunteers will participate in two visits: (1) Visit 1, baseline and (2) Visit 2, follow up. At each visit, volunteers will report to the Olin Physical Lab room 208 after having fasted for 3 hours prior. They can drink water one hour before the visit. Participants will be instructed not to use anti-bacterial mouthwash the day of the visit. The participant will be asked to provide 4 mL of saliva and a study team member will collect a bacterial sample from the posterior dorsal surface of their tongue (as described below). These samples will be frozen at -80 degrees for genetic analysis and identification of bacterial strains.

After saliva and tongue samples are collected, blood will be drawn (as described below) for plasma nitrite and nitrate determination. This blood sample will be the "pre-" sample collected at baseline and follow-up. Volunteers will then drink one 70 mL Beet it Sport Nitrate 400 shot (https://www.beet-it.us/pages/beet-it-sports). A "post-" blood draw will be collected 2.5 hours after consumption of the beetroot juice.

At Visit 1, after the second blood draw, volunteers will receive 7 days worth of either probiotic or the placebo. Volunteers will consume the probiotic (or placebo) as indicated by the manufacturer of the probiotic once a day. On day 8, the volunteers will return for visit 2.

The data will include (1) baseline and follow-up analysis of oral bacterial strains and (2) Pre- and post-beet juice consumption plasma nitrite and nitrate levels. The investigators hypothesize that the abundance of Lactobacillus will be higher at follow-up compared to baseline for volunteers taking the probiotic but that there will be no change in the placebo group. The investigators also hypothesize that the change in plasma nitrite (post minus pre) will be lower at follow-up than at baseline for volunteers taking the probiotic but that there will be no change in the placebo group.

* Study Materials (all commercially available):

  1. Placebo: Honest Placebo Pills by Zeebo
  2. Herbiotics Oral + Ent Probiotic
  3. Beet it Sport Nitrate 400 shot
* Collection of Saliva and Tongue scraping. Volunteers will report to the Olin Physical Lab room 208 after having fasted for 3 hours prior. They can drink water one hour before the visit. Participants will be instructed not to use anti-bacterial mouthwash the day of the visit. The participant will be asked to provide 4 mL of saliva by spitting into a microcentrifuge tube. For the tongue samples, a HydraFlock 6" Sterile Large Flock Swab w/Polystyrene Handle (Puritan Medical) will be used to collect scrapings. Volunteers will be asked to open their mouths as wide as possible and stick out their tongue. The posterior 1/3 of the dorsal surface of the tongue will be sampled by scraping lightly to moderately firmly the dorsal surface of the tongue back and forth Scraping will take a minute or so. The tongue scraping will be placed in 0.85 mL of buffered sterile saline and 0.15 mL glycerol. All samples will be frozen at -80°C and sent to Professor Hariom Yadav at the University of South Florida for genomic analysis.
* Blood draws and processing Blood will be drawn by a certified, trained phlebotomist. Blood samples (maximum ~10 mL) will be collected from participants following consent. Blood will be collected at each visit pre and 2.5 hours post beet juice consumption. Blood will be drawn as close to the 2.5 hour mark as possible. Realistically, it may occur between 2 to 3 hours after the final study beverage is consumed. Blood will be drawn by lab personnel with certified phlebotomy training via standard venipuncture methods or Tasso HemolinkTM device. The HemoLinkTM is an FDA-approved blood collection device that uses small lancets and gentle suction to collect a very small sample (~ ¼ teaspoons) of blood. Blood will be collected in standard blood collection tubes (e.g. citrate (blue-top), EDTA (purple-top) and heparin (green-top)) and labeled appropriately. The preferred tube is a 4 mL heparin tube. All blood samples drawn for research purposes will be identified by the study participant number and date/time of collection, which will also be recorded on the standardized data collection form. No personal identifying information will be included on the samples processed for research purposes. All blood samples will be immediately spun immediately in a centrifuge at 600-800g for five minutes and the supernatant collected. The plasma will be frozen on dry ice and then stored at -80°C for analysis of nitrite and nitrate content.
* Probiotic or placebo consumption Both the probiotic and placebo will be consumed twice a day according to instructions for the probiotic. One capsule is chewed or allowed to melt in the volunteer's mouth and then the contents are switched around in the mouth before being swallowed.

Risks Approximately 10 mL of blood will be drawn from patients willing to participate. This will be done in the usual fashion, preparing the venipuncture site with the local anesthetic EMLA, then drawing blood through a small gauge (23 or 21) butterfly needle. Drawing blood from a vein may be associated with discomfort or bruising at the site of needle puncture. Rarely, fainting or infection at the site of needle puncture may occur. All blood will be drawn from a person trained in phlebotomy. There will be no way to trace the blood back to the donor.

There are no known health risks for donating saliva or tongue scrapings from individuals who will be included in the study. There is a very minimal risk of linking individuals to the study. There will be no way to trace the saliva or tongue scrapings back to the donor.

Protections Against Risk Strategies for protection against risk. To protect privacy of participants and confidentiality of research data, no personal information regarding individual participants will be linked to the in vitro studies.

Plans for medical attention. In case of injury (which is extremely unlikely) as a result of saliva donation, the individuals will be instructed to contact their physician and medical care will be offered and charged to available research coverage maintained at Wake Forest School of Medicine.

In case of injury as a result of blood drawing, the patients will be instructed to contact their physician and medical care will be offered and charged to available research coverage maintained at Wake Forest School of Medicine. Blood drawn on the Reynolda campus is not a clinical setting, but blood will be drawn by trained phlebotomists with years of experience who maintain their training.

Any unanticipated problems, serious and unexpected adverse events, deviations or protocol changes will be promptly reported by the principal investigator or designated member of the research team to the IRB and sponsor or appropriate government agency if appropriate.

Incidental Findings. No incidental findings are expected to be discovered in this study as measures of bacterial nitrate reduction are not currently of clinical relevance so a strange, individual result in that measure would not be worth communicating.

Sample size assessment and statistical analysis

The investigators plan to enroll 10 participants who receive the probiotic and 10 participants who receive the placebo. The investigators hypothesize that, using a paired t-test, participants taking the probiotic will have significantly (P < .05) lower change in plasma nitrite (post minus pre) at follow up compared to baseline while there will be no significant effect of the placebo (paired t-test).

The Investigators calculated that they would have 80% power to measure a 75% decrease in the change in nitrite at follow-up compared to baseline for the probiotic group with 10 participants per group (Continuous endpoint Two independent samples). The investigators assumed a 60% standard deviation in the change in nitrite for follow-up vs baseline based on previous data from our lab.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers ages 18-70

Exclusion Criteria:

* Individuals with a history of difficult blood draws. More than 2 blood draws in one week; on anti-coagulant or anti-platelet therapy (e.g. aspirin, Coumadin, etc.); known pregnancy; in police custody or a prisoner; common illness within 2 weeks of potential enrollment. The cumulative volume of blood drawn from a healthy adult over the prior eight-week period would exceed 550 ml including the current draw.
* In addition, individuals uncomfortable spitting into a tube, dry mouth (xerostomia) or dry eyes, Patients suffering from autoimmune diseases such as Sjogren's syndrome, rheumatoid arthritis, systemic lupus erythematosus, or progressive systemic sclerosis, since individuals with these autoimmune inflammatory diseases exhibit persistent xerostomia, individuals with active caries diagnosis or history of periodontitis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Dietary Nitrate Conversion to Plasma Nitrite | The two visits will be 8 days apart.
  The main outcome is the plasma nitrite level 2.5 after consuming Beet Juice minus the plasma nitrite level prior to drinking beet juice. Blood will be collected prior to drinking one Beet it Sport shot and 2.5 hours after drinking the shot. Plasma nitrite will be measured from these blood draws.
  This outcome will be measured at two visits: baseline and followup (day 8) and the increase in plasma nitrite at the two visits will be compared. Between the two visits the participants will consume the Probiotic or Placebo for 7 days.

SECONDARY OUTCOMES:
Percentage Lactobacillus | The two visits will be 8 days apart.
  Oral bacterial species will be determined from saliva and tongue scrapings at both visits prior to beet juice consumption. The percentage abundance of Lactobacillus will be determined at each visit and compared to each other. Between the two visits the participants will consume the Probiotic or Placebo for 7 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Wake Forest University, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Only a coded participant identifier will be shared with a scientific collaborator. The participant identifier will not be traceable to the individual participant. It is only used to correlate data collected at different sites.
Supporting Information: Analytic Code
Time Frame: When saliva and tongue scrapings are sent to University of South Florida for microbiome analysis, the samples will include the code.
Access Criteria: Scientific investigators on the team will have access to the codes - not any links to the original participants.

REFERENCES:
- [Background] Leiva A, Fuenzalida B, Barros E, Sobrevia B, Salsoso R, Saez T, Villalobos R, Silva L, Chiarello I, Toledo F, Gutierrez J, Sanhueza C, Pardo F, Sobrevia L. Nitric Oxide is a Central Common Metabolite in Vascular Dysfunction Associated with Diseases of Human Pregnancy. Curr Vasc Pharmacol. 2016;14(3):237-59. doi: 10.2174/1570161114666160222115158. PMID 26899560
- [Background] Almeida CB, Souza LE, Leonardo FC, Costa FT, Werneck CC, Covas DT, Costa FF, Conran N. Acute hemolytic vascular inflammatory processes are prevented by nitric oxide replacement or a single dose of hydroxyurea. Blood. 2015 Aug 6;126(6):711-20. doi: 10.1182/blood-2014-12-616250. Epub 2015 May 27. PMID 26019278
- [Background] Maley JH, Lasker GF, Kadowitz PJ. Nitric oxide and disorders of the erythrocyte: emerging roles and therapeutic targets. Cardiovasc Hematol Disord Drug Targets. 2010 Dec 1;10(4):284-91. doi: 10.2174/187152910793743878. PMID 21067512
- [Background] Eisenhut M. Severe hemolysis as a potential contributing factor in the pathophysiology of cerebral malaria. Clin Infect Dis. 2015 Apr 1;60(7):1138. doi: 10.1093/cid/ciu1149. Epub 2014 Dec 19. No abstract available. PMID 25527655
- [Background] Donadee C, Raat NJ, Kanias T, Tejero J, Lee JS, Kelley EE, Zhao X, Liu C, Reynolds H, Azarov I, Frizzell S, Meyer EM, Donnenberg AD, Qu L, Triulzi D, Kim-Shapiro DB, Gladwin MT. Nitric oxide scavenging by red blood cell microparticles and cell-free hemoglobin as a mechanism for the red cell storage lesion. Circulation. 2011 Jul 26;124(4):465-76. doi: 10.1161/CIRCULATIONAHA.110.008698. Epub 2011 Jul 11. PMID 21747051
- [Background] Gladwin MT, Kim-Shapiro DB. Storage lesion in banked blood due to hemolysis-dependent disruption of nitric oxide homeostasis. Curr Opin Hematol. 2009 Nov;16(6):515-23. doi: 10.1097/MOH.0b013e32833157f4. PMID 19701085
- [Background] Hirai DM, Musch TI, Poole DC. Exercise training in chronic heart failure: improving skeletal muscle O2 transport and utilization. Am J Physiol Heart Circ Physiol. 2015 Nov;309(9):H1419-39. doi: 10.1152/ajpheart.00469.2015. Epub 2015 Aug 28. PMID 26320036
- [Background] Voetsch B, Jin RC, Loscalzo J. Nitric oxide insufficiency and atherothrombosis. Histochem Cell Biol. 2004 Oct;122(4):353-67. doi: 10.1007/s00418-004-0675-z. Epub 2004 Aug 26. PMID 15338226
- [Background] Bertoluci MC, Ce GV, da Silva AM, Wainstein MV, Boff W, Punales M. Endothelial dysfunction as a predictor of cardiovascular disease in type 1 diabetes. World J Diabetes. 2015 Jun 10;6(5):679-92. doi: 10.4239/wjd.v6.i5.679. PMID 26069717
- [Background] Kapil V, Haydar SM, Pearl V, Lundberg JO, Weitzberg E, Ahluwalia A. Physiological role for nitrate-reducing oral bacteria in blood pressure control. Free Radic Biol Med. 2013 Feb;55:93-100. doi: 10.1016/j.freeradbiomed.2012.11.013. Epub 2012 Nov 23. PMID 23183324
- [Background] Govoni M, Jansson EA, Weitzberg E, Lundberg JO. The increase in plasma nitrite after a dietary nitrate load is markedly attenuated by an antibacterial mouthwash. Nitric Oxide. 2008 Dec;19(4):333-7. doi: 10.1016/j.niox.2008.08.003. Epub 2008 Aug 30. PMID 18793740
- [Background] Webb AJ, Patel N, Loukogeorgakis S, Okorie M, Aboud Z, Misra S, Rashid R, Miall P, Deanfield J, Benjamin N, MacAllister R, Hobbs AJ, Ahluwalia A. Acute blood pressure lowering, vasoprotective, and antiplatelet properties of dietary nitrate via bioconversion to nitrite. Hypertension. 2008 Mar;51(3):784-90. doi: 10.1161/HYPERTENSIONAHA.107.103523. Epub 2008 Feb 4. PMID 18250365
- [Background] Lundberg JO, Weitzberg E, Gladwin MT. The nitrate-nitrite-nitric oxide pathway in physiology and therapeutics. Nat Rev Drug Discov. 2008 Feb;7(2):156-67. doi: 10.1038/nrd2466. PMID 18167491
- [Background] Helms CC, Liu X, Kim-Shapiro DB. Recent insights into nitrite signaling processes in blood. Biol Chem. 2017 Mar;398(3):319-329. doi: 10.1515/hsz-2016-0263. PMID 27611767
- [Background] DeMartino AW, Kim-Shapiro DB, Patel RP, Gladwin MT. Nitrite and nitrate chemical biology and signalling. Br J Pharmacol. 2019 Jan;176(2):228-245. doi: 10.1111/bph.14484. Epub 2018 Oct 3. PMID 30152056
- [Background] Presley TD, Perlegas AS, Bain LE, Ballas SK, Nichols JS, Sabio H, Gladwin MT, Kato GJ, Kim-Shapiro DB. Effects of a single sickling event on the mechanical fragility of sickle cell trait erythrocytes. Hemoglobin. 2010;34(1):24-36. doi: 10.3109/03630260903546999. PMID 20113285
- [Background] Eggebeen J, Kim-Shapiro DB, Haykowsky M, Morgan TM, Basu S, Brubaker P, Rejeski J, Kitzman DW. One Week of Daily Dosing With Beetroot Juice Improves Submaximal Endurance and Blood Pressure in Older Patients With Heart Failure and Preserved Ejection Fraction. JACC Heart Fail. 2016 Jun;4(6):428-37. doi: 10.1016/j.jchf.2015.12.013. Epub 2016 Feb 10. PMID 26874390
- [Background] Petrie M, Rejeski WJ, Basu S, Laurienti PJ, Marsh AP, Norris JL, Kim-Shapiro DB, Burdette JH. Beet Root Juice: An Ergogenic Aid for Exercise and the Aging Brain. J Gerontol A Biol Sci Med Sci. 2017 Sep 1;72(9):1284-1289. doi: 10.1093/gerona/glw219. PMID 28329785
- [Background] Larsen FJ, Weitzberg E, Lundberg JO, Ekblom B. Dietary nitrate reduces maximal oxygen consumption while maintaining work performance in maximal exercise. Free Radic Biol Med. 2010 Jan 15;48(2):342-7. doi: 10.1016/j.freeradbiomed.2009.11.006. Epub 2009 Nov 12. PMID 19913611
- [Background] Kapil V, Khambata RS, Robertson A, Caulfield MJ, Ahluwalia A. Dietary nitrate provides sustained blood pressure lowering in hypertensive patients: a randomized, phase 2, double-blind, placebo-controlled study. Hypertension. 2015 Feb;65(2):320-7. doi: 10.1161/HYPERTENSIONAHA.114.04675. Epub 2014 Nov 24. PMID 25421976
- [Background] Velmurugan S, Kapil V, Ghosh SM, Davies S, McKnight A, Aboud Z, Khambata RS, Webb AJ, Poole A, Ahluwalia A. Antiplatelet effects of dietary nitrate in healthy volunteers: involvement of cGMP and influence of sex. Free Radic Biol Med. 2013 Dec;65:1521-1532. doi: 10.1016/j.freeradbiomed.2013.06.031. Epub 2013 Jun 24. PMID 23806384
- [Background] Velmurugan S, Gan JM, Rathod KS, Khambata RS, Ghosh SM, Hartley A, Van Eijl S, Sagi-Kiss V, Chowdhury TA, Curtis M, Kuhnle GG, Wade WG, Ahluwalia A. Dietary nitrate improves vascular function in patients with hypercholesterolemia: a randomized, double-blind, placebo-controlled study. Am J Clin Nutr. 2016 Jan;103(1):25-38. doi: 10.3945/ajcn.115.116244. Epub 2015 Nov 25. PMID 26607938
- [Background] Kerley CP, Cahill K, Bolger K, McGowan A, Burke C, Faul J, Cormican L. Dietary nitrate supplementation in COPD: an acute, double-blind, randomized, placebo-controlled, crossover trial. Nitric Oxide. 2015 Jan 30;44:105-11. doi: 10.1016/j.niox.2014.12.010. Epub 2014 Dec 19. PMID 25534960
- [Background] Kerley CP, O'Neill JO, Reddy Bijjam V, Blaine C, James PE, Cormican L. Dietary nitrate increases exercise tolerance in patients with non-ischemic, dilated cardiomyopathy-a double-blind, randomized, placebo-controlled, crossover trial. J Heart Lung Transplant. 2016 Jul;35(7):922-6. doi: 10.1016/j.healun.2016.01.018. Epub 2016 Jan 16. No abstract available. PMID 27009674
- [Background] Shaltout HA, Eggebeen J, Marsh AP, Brubaker PH, Laurienti PJ, Burdette JH, Basu S, Morgan A, Dos Santos PC, Norris JL, Morgan TM, Miller GD, Rejeski WJ, Hawfield AT, Diz DI, Becton JT, Kim-Shapiro DB, Kitzman DW. Effects of supervised exercise and dietary nitrate in older adults with controlled hypertension and/or heart failure with preserved ejection fraction. Nitric Oxide. 2017 Sep 30;69:78-90. doi: 10.1016/j.niox.2017.05.005. Epub 2017 May 23. PMID 28549665
- [Background] Wilkerson DP, Hayward GM, Bailey SJ, Vanhatalo A, Blackwell JR, Jones AM. Influence of acute dietary nitrate supplementation on 50 mile time trial performance in well-trained cyclists. Eur J Appl Physiol. 2012 Dec;112(12):4127-34. doi: 10.1007/s00421-012-2397-6. Epub 2012 Apr 20. PMID 22526247
- [Background] Kenjale AA, Ham KL, Stabler T, Robbins JL, Johnson JL, Vanbruggen M, Privette G, Yim E, Kraus WE, Allen JD. Dietary nitrate supplementation enhances exercise performance in peripheral arterial disease. J Appl Physiol (1985). 2011 Jun;110(6):1582-91. doi: 10.1152/japplphysiol.00071.2011. Epub 2011 Mar 31. PMID 21454745
- [Background] Ormesher L, Myers JE, Chmiel C, Wareing M, Greenwood SL, Tropea T, Lundberg JO, Weitzberg E, Nihlen C, Sibley CP, Johnstone ED, Cottrell EC. Effects of dietary nitrate supplementation, from beetroot juice, on blood pressure in hypertensive pregnant women: A randomised, double-blind, placebo-controlled feasibility trial. Nitric Oxide. 2018 Nov 1;80:37-44. doi: 10.1016/j.niox.2018.08.004. Epub 2018 Aug 9. PMID 30099096
- [Background] Hyde ER, Andrade F, Vaksman Z, Parthasarathy K, Jiang H, Parthasarathy DK, Torregrossa AC, Tribble G, Kaplan HB, Petrosino JF, Bryan NS. Metagenomic analysis of nitrate-reducing bacteria in the oral cavity: implications for nitric oxide homeostasis. PLoS One. 2014 Mar 26;9(3):e88645. doi: 10.1371/journal.pone.0088645. eCollection 2014. PMID 24670812
- [Background] Rosier BT, Moya-Gonzalvez EM, Corell-Escuin P, Mira A. Isolation and Characterization of Nitrate-Reducing Bacteria as Potential Probiotics for Oral and Systemic Health. Front Microbiol. 2020 Sep 15;11:555465. doi: 10.3389/fmicb.2020.555465. eCollection 2020. PMID 33042063